CLINICAL TRIAL: NCT05584553
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the ToggleLoc™ 2.9mm and the JuggerLoc™ Soft Tissue Systems (Implants and Instrumentation) in the Shoulder - A Multicenter Retrospective Study
Brief Title: PMCF Study on the Safety, Performance and Clinical Benefits Data of the ToggleLoc™ 2.9mm and JuggerLoc™ in the Shoulder
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-70SM
Record Dates: First submitted 2022-04-25; First posted 2022-10-18 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-12

CONDITIONS: Bankart Lesions; SLAP Lesion; Acromioclavicular; Dislocation; Capsular Shift/Capsulolabral Reconstruction; Deltoid Repair; Rotator Cuff Tear Repair; Biceps Tendon Disorder
Keywords: Post-Market Clinical Follow-Up Study; Medical Device; Performance; Safety; Clinical Benefits
MeSH Terms: conditions — Bankart Lesions; Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- ToggleLoc 2.9 mm soft tissue device: Patients who already received the ToggleLoc 2.9 mm soft tissue device in the shoulder. No additional surgery will be performed.
  Interventions: Device: ToggleLoc 2.9 mm soft tissue device
- JuggerLoc soft tissue device: Patients who already received the JuggerLoc soft tissue device in the shoulder. No additional surgery will be performed.
  Interventions: Device: JuggerLoc soft tissue device

INTERVENTIONS:
Device: ToggleLoc 2.9 mm soft tissue device — The ToggleLoc 2.9 mm Soft Tissue devices consist of non-resorbable devices intended to aid in arthroscopic and orthopaedic reconstructive procedures requiring soft tissue to bone fixation.
  Groups: ToggleLoc 2.9 mm soft tissue device
Device: JuggerLoc soft tissue device — The JuggerLoc Soft Tissue devices consist of non-resorbable devices intended to aid in arthroscopic and orthopaedic reconstructive procedures requiring soft tissue to bone fixation.
  Groups: JuggerLoc soft tissue device

SUMMARY:
The study is a multicenter, retrospective, non-randomized, non-controlled and consecutive series post-market study. The purpose of this study is to collect data confirming safety, performance and clinical benefits of the ToggleLoc 2.9 mm and the JuggerLoc Soft Tissue Systems when used for soft tissue to bone fixation in the shoulder.

The primary objective is the assessment of performance by analyzing soft tissue to bone healing in the shoulder.

The secondary objective is the assessment of safety and clinical benefits. Safety will be evaluated by recording and analyzing the incidence and frequency of complications and adverse events. Relation of the events to device, instrumentation and/or procedure will be specified. Clinical benefits will be assessed by recording patient-reported outcome measures (PROMs) at the longest follow-up after surgery (minimum one year).

DETAILED DESCRIPTION:
The ToggleLoc 2.9 mm and JuggerLoc Soft Tissue devices consist of non-resorbable devices intended to aid in arthroscopic and orthopaedic reconstructive procedures requiring soft tissue to bone fixation. The clinical purpose is to restore the function and flexibility of the shoulder requiring soft tissue to bone fixation and to relieve pain that cannot be controlled by other treatments.

Three sites will be involved in this study. The aim is to include a total of 206 (103 cases operated with the ToggleLoc 2.9 mm and 103 cases operated with the JuggerLoc in the shoulder) consecutive series cases. All potential study subjects will be required to participate in the Informed Consent Process.

Baseline data from the preop and intraop will be available in medical notes. The patients will be asked to complete patient questionnaires during a minimum 1 year follow up visit/phone call. In addition, any complications and adverse events that occured since the surgery will also be collected during the follow-up visit/phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patients that received the ToggleLoc 2.9 mm and/or the JuggerLoc Soft Tissue devices for soft tissue to bone fixation in the shoulder.
* Patients 18 years or older and skeletally mature.
* Patients capable of understanding the surgeon's explanations and following his/her instructions, able and willing to participate in the follow-up program and who gave consent to take part in the study.

Exclusion Criteria:

* Infection.
* Patient conditions including blood supply limitations, and insufficient quantity or quality of bone or soft tissue.
* Patients with mental or neurologic conditions who are unwilling or incapable of following postoperative care instructions.
* Foreign body sensitivity. Where material sensitivity is suspected, testing is to be completed prior to implantation of the device.
* Patients who are unwilling or unable to give consent, or to comply with the follow-up program.
* Patients who have any condition that would in the judgment of the Investigator place the patient at undue risk or interfere with the study.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant).
* Off-label use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had required a soft tissue to bone fixation in the shoulder with the ToggleLoc 2.9 mm and/or the JuggerLoc Soft Tissue devices according to Zimmer Biomet's Instruction for Use (IFU) and and who meet all the inclusions criteria and none of the exclusions criteria.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan ACHAKRI, Study Director — Zimmer Biomet
Locations (3):
- Advanced Bone and Joint, City of Saint Peters, Missouri, United States
- Spain (2):
  - Centro Médico Quirónsalud, Alicante
  - Hospital Universitario Quirónsalud, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device | JuggerLoc Soft Tissue Device
Started | 106 | 108
Completed | 106 | 108
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device | JuggerLoc Soft Tissue Device | Total
Number analyzed (Participants) | 106 | 108 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 95 | 192
  >=65 years | 9 | 13 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.7 (9.0) | 47.1 (11.3) | 50.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 80 | 84 | 164
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 40 | 120
  Spain | 26 | 68 | 94
Body Mass Index of participants [Mean (Standard Deviation); unit: kg/m²] | 30.1 (5.6) | 29.1 (5.1) | 29.5 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Evidence of Soft Tissue-to-Bone Healing in the Shoulder
Description: Assessment of performance by analyzing soft tissue to bone healing in the shoulder. The principal investigator will clinically evaluate the study shoulder to assess if soft tissue to bone healing has occurred using an assessment of pain. Healing was assessed by clinical examination at a minimum of 12 months post-operation. Soft tissue-to-bone healing was evaluated through clinical assessment at follow-up. Healing was defined as restoration of tendon attachment to bone without visible gap, pain, or functional limitation. Clinical evaluation included absence of pain on palpation and a satisfactory range of motion. Results represent the number of participants meeting these criteria for complete healing.
Time Frame: From operation to the study completion, minimum 1 year post-op. Through last available follow-up (mean = 2.1 years, range = 1.0-5.2 years for JuggerLoc; mean = 3.5 years, range = 1.0-7.0 years for ToggleLoc)
Measure: Number; unit: participants
Units Other Than Participants: Implants
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device | JuggerLoc Soft Tissue Device
Number analyzed (Participants) | 106 | 108
Number analyzed (Implants) | 106 | 108
participants | 106 | 108

2. Secondary Outcome: Number of Participants With Revision Surgery
Description: Safety will be evaluated by recording and analyzing the incidence of revisions. A Kaplan-Meier survival curve will be calculated. Revisions were defined as any subsequent surgical intervention involving removal, replacement, or modification of the index implant. Data were analyzed descriptively and using Kaplan-Meier survival analysis to estimate the probability of remaining revision-free over time. Results represent the number of participants who underwent at least one revision during follow-up.
Time Frame: From date of surgery to last available follow-up (mean follow-up = 2.1 ± 1.1 years for JuggerLoc and 3.5 ± 2.0 years for ToggleLoc), minimum 1 year post-op.
Measure: Count of Participants; unit: Participants
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device | JuggerLoc Soft Tissue Device
Number analyzed (Participants) | 106 | 108
Participants | 0 | 0

3. Secondary Outcome: EuroQol Five-dimensional Health Questionnaire (EQ-5D-5L)
Description: Clinical benefits will be assessed by recording patient-reported outcome measures (PROMs). This standardized instrument includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The EQ-5D is a standardized instrument widely used to measure health status. It is a self-reported assessment about the patient's quality of life composed of two parts: a questionnaire and a visual analogue scale (VAS). The questionnaire includes 5 questions referring to mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each question can be answered in five ways, indicating no, slight, moderate, severe problems or inability to complete the task. In the derived EQ-5D-5L score, the highest score is 1 and the lowest score is -0.573; negative numbers correspond to a self-assessed health state. The VAS is a vertical scale ranging from 100 ('The best health you can imagine') to 0 ('The worst health you can imagine').
Time Frame: From pre-operative baseline to last available follow-up (mean follow-up = 2.1 ± 1.1 years for JuggerLoc and 3.5 ± 2.0 years for ToggleLoc). Minimum 1 year post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device | JuggerLoc Soft Tissue Device
Number analyzed (Participants) | 106 | 108
score on a scale | 79.6 (16.2) | 84.9 (10.9)

4. Secondary Outcome: Oxford Shoulder Score (OSS)
Description: Clinical benefits will be assessed by recording patient-reported outcome measures (PROMs). The Oxford Shoulder Score (OSS) is a patient-reported outcome questionnaire that was developed to specifically assess the patient's perspective of outcome following shoulder arthroplasty. The OSS consists of twelve questions covering function and pain. To calculate the total score, each question is scored from 0 (worst outcome) to 4 (best outcome), and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The outcome score can be categorized as: Satisfactory Joint Function: 40 - 48, Moderate-Mild Arthritis: 30 - 39, Moderate-Severe Arthritis: 20 - 29, Severe Arthritis: 0 - 19.
Time Frame: From pre-operative baseline to last available follow-up (mean follow-up = 2.1 ± 1.1 years for JuggerLoc and 3.5 ± 2.0 years for ToggleLoc), minimum 1 year post-op.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device | JuggerLoc Soft Tissue Device
Number analyzed (Participants) | 106 | 108
score on a scale | 45.4 (5.4) | 45.5 (5.0)

ADVERSE EVENTS:
Time Frame: From date of surgery to last available follow-up (mean = 2.1 ± 1.1 years for the JuggerLoc arm and 3.5 ± 2.0 years for the ToggleLoc arm)
Description: Adverse events were prospectively collected using the Oracle RDC electronic data-capture system. For each event, the date of occurrence, event type, relationship to the study device, treatment provided, and treatment outcome were recorded.
Arm/Group | ToggleLoc 2.9 mm Soft Tissue Device | JuggerLoc Soft Tissue Device
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/106 | 1/108
Other Adverse Events (participants affected / at risk) | 23/106 | 1/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ToggleLoc 2.9 mm Soft Tissue Device (N=106) | JuggerLoc Soft Tissue Device (N=108)
GULLIAN BARRE SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) — PATIENT DIAGNOSED WITH GULLIAN BARRE SYNDROME. WAS HOSPILIZED 84 DAYS. CURRENTLY IN REHAB. SHOULDER IS DOING GREAT
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ToggleLoc 2.9 mm Soft Tissue Device (N=106) | JuggerLoc Soft Tissue Device (N=108)
SEVERE BLISTERING FROM THE TAPE. (Skin and subcutaneous tissue disorders) | 0 (0) | 1/1 (1) — 2 DAYS POST OP [ PATIENT HAD "SEVERE" BLISTERING FROM THE TAPE. IT RESOLVED BUT HAS SCARRING
Urinary (Renal and urinary disorders) | 1 (1) | 0 (0) — PATIENT RECALLS NOT BEING ABLE TO URINATE. WENT TO THE ED AND CATHETER WAS PLACED. PCP EVENTUALLY REMOVED.
Bleeding (Surgical and medical procedures) | 1 (1) | 0 (0) — PATIENT CAME IN POD 1 WITH BLEEDING CONCERNS. NO ACTIVE BLEEDING. NEW DRESSING APPLIED. POST OP VISIT: THE INCISION LOOKED FINE
Bleeding (Surgical and medical procedures) | 1 (1) | 0 (0) — PATIENT CAME INTO THE OFFICE FOR EARLY FOLLOW UP FOR BLEEDING CONCERNS. NO ACTIVE BLEEDING. DRESSING REAPPLIED
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) — PATIENT RECALLS CHEST PAIN AND ADMITTED THRU ED. H/O 1992 STENTING AND MI. 1/31/18 OFFICE NOTE STATES HE SAW CARDIOLOGY AND WAS GETTING A WORK UP THAT DAY. .
Bicep Pain (Nervous system disorders) | 1 (1) | 0 (0) — POST OP VISIT PATIENT MENTIONS N/T AROUND BICEP INCISION. NO MENTION AT FUTURE APPTS.
Knee Injection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — SEEN FOR 3RD RIGHT KNEE EUFLEXXA INJECTION (FIRST TWO PRIOR INJECTIONS GIVEN PRIOR TO SHOULDER SURGERY.)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — POST OP VISIT PATIENT HAD A RASH UNDER OPERATED ARM
Small Wound (Infections and infestations) | 1 (1) | 0 (0) — SMALL WOUND DEHISCENCE WHICH REQUIRED ANTIBIOTICS
Neck, Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — EARLY FOLLOW UP DUE TO NECK, MID-BACL, AND SCAPULA PAIN THAT STARTED A FEW DAYS
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — FOLLOW UP: STATES PATIENT IS DOING STROKE REHAB.
LATERAL EPICONDYLITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — REPORTS NUMBNESS IN FOREARM AND ELBOW PAIN. LATERAL EPICONDYLITIS- NO ADDITIONAL TREATMENT
RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient HAVING RIGHT SHOULDER PAIN-REPORTS "LONG HISTORY" OF RIGHT SHOULDER PAIN- SHOULDER XRAY AND EVALUATED BUT PATIENT DIDNT WANT FUTHUR TREATMENT
Pain (General disorders) | 1 (1) | 0 (0) — THE PATIENT HAD INCREASED PAIN AFTER WORKING OUT. WENT TO PT. DID GET BETTER. NORMAL EXAM
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — RIGHT SHOULDER PAIN - NON Study Related
Left Hand Pain (Nervous system disorders) | 1 (1) | 0 (0) — Left Hand Pain (non study related) - Patient doesn't want to Follow up
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Hip Pain - Resolved
Patient Fell (General disorders) | 1 (1) | 0 (0) — PATIENT FELL ON LEFT SIDE GETTING INTO A VAN
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient experienced pain in left hand - Diagnosed with Carpal tunnel syndrome
Hand Pain (Nervous system disorders) | 1 (1) | 0 (0) — HAND PAIN. INJECTION GIVEN LEFT HAND. Resolved
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Knee Pain - Injections, resolved
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — NON DISPLACED ANKLE FRACTURE. NON OPERATIVE TREATMENT
PAIN (Nervous system disorders) | 1 (1) | 0 (0) — PERSISTANCE PAIN (NON STUDY RELATED), INJECTION. DEPO MEDROL 40MG AND 1% LIDOCAINE
Injury (General disorders) | 1 (1) | 0 (0) — REPORTS INJURY WHEN GRABBING A DOOR WEEKS AGO. HAD INCREASED PAIN. IMPROVED OVER LAST FEW WEEKS

LIMITATIONS AND CAVEATS:
The retrospective setting of the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT05584553/Prot_SAP_000.pdf